CLINICAL TRIAL: NCT00561457
Title: A Clinical Evaluation of the Bard® Luminexx™ Iliac Stent and Delivery System
Acronym: Luminexx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-1021
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Iliac Artery Occlusive Disease
Keywords: Iliac; Artery; Occlusive; Stenosis
MeSH Terms: conditions — Bites and Stings; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iliac Stenting (Experimental): Stent placement in the iliac artery
  Interventions: Device: Bard Luminexx Iliac Stent and Delivery System

INTERVENTIONS:
Device: Bard Luminexx Iliac Stent and Delivery System — Iliac Stenting

SUMMARY:
To determine the safety and effectiveness of the LUMINEXX stent for the proposed indication of treatment of common and/or external iliac artery occlusive disease

DETAILED DESCRIPTION:
The study is designed to collect safety and efficacy data on the Bard Luminexx Iliac Stent in a broad patient population having indications for iliac stenting. Effectiveness in this study will be demonstrated by the prevention of Major Adverse Clinical Events (MACE). The composite primary endpoint of this clinical trial is freedom from peri-procedural death and freedom from stented segment revascularization or restenosis (>50%) at nine months.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legal guardian understands procedure and provides written informed consent prior to study participation.
* Patient must be able and willing to comply with all study procedures including scheduled follow-up visits and diagnostic tests.
* Lesion(s) distinctly localized in the common and/or external iliac arteries.
* Reference lumen diameter (RLD) 6 mm and 9 mm.
* Stenosis 30% and symptomatic ischemic disease (Category 1-6 Chronic Limb Ischemia or Threatened or Irreversible Acute Limb Ischemia).

Exclusion Criteria:

* Patients diagnosed with preoperative coagulation disorder or with contraindications to antiplatelet or anticoagulant therapy.
* Patients who are pregnant or planning to become pregnant during the clinical investigation.
* Patients with a life expectancy < 3 years.
* Patients currently or scheduled to be enrolled in another investigation that conflicts with follow-up testing or may confound the study data.
* Patients with absolute contraindication to x-ray contrast media or medications normally administered during an interventional procedure.
* Patients with severe tortuosity or angulation of a vessel that may prevent access in the opinion of the investigator.
* The presence of soft, thrombotic or embolic material within or adjacent to the lesion(s) being treated with the study device, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2003-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment was completed November 1, 2004 with a total of 134 patients from 9 study sites.
Groups:
- Luminexx Iliac Stent and Delivery System: Bard® LUMINEXX* Iliac Stent and the Bard® LUMINEXX* 6F Iliac Stent systems.
Period: Overall Study
Arm/Group | Luminexx Iliac Stent and Delivery System
Started | 134
Completed | 110
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Luminexx Iliac Stent and Delivery System
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.31 (10.31)
Gender [Count of Participants; unit: Participants]
  Female | 61
  Male | 73
Region of Enrollment [Number; unit: participants]
  United States | 134

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major Adverse Clinical Events (MACE)
Description: Major Adverse Clinical Events defined as peri-procedural death (death during the procedure or prior to hospital discharge), target lesion revascularization (TLR), or stented segment restenosis (> 50%) at nine months postprocedure.
Time Frame: 9-months
Population: The analysis was an intention to treat (ITT)population which included the data for all completed patients (those who had a MACE event within 9-months and those who reached 9 months without experiencing an event). Natural censoring was used in the analysis according to the statistical analysis plan.
Measure: Mean (95% Confidence Interval); unit: MACE events per 9 months
Arm/Group | Luminexx Iliac Stent and Delivery System
Number analyzed (Participants) | 110
MACE events per 9 months | 0.153 [0.0905 to 0.2292]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Luminexx Iliac Stent and Delivery System
Serious Adverse Events (participants affected / at risk) | 57/134
Other Adverse Events (participants affected / at risk) | 13/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luminexx Iliac Stent and Delivery System (N=134)
Distal Revascularization (Target Limb) (Surgical and medical procedures) | 16 (25)
Revascularization (Non-target Limb) (Surgical and medical procedures) | 13 (14)
Bleeding (Vascular disorders) | 6 (6)
Angina/Coronary Ischemia (Cardiac disorders) | 9 (9)
Sepsis (Vascular disorders) | 6 (8)
Arterial Thrombosis (Vascular disorders) | 5 (8)
Target Lesion Revascularization (Surgical and medical procedures) | 2 (2)
False Aneurysm (Injury, poisoning and procedural complications) | 4 (4)
Amputation on Study Side Limb (Surgical and medical procedures) | 4 (4)
Arrhythmia (Cardiac disorders) | 5 (8)
Sudden Cardiac Death (Cardiac disorders) | 2 (2)
Stroke (Nervous system disorders) | 4 (4)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Carotid Artery Disease (Nervous system disorders) | 4 (4)
Congestive Heart Failure (Cardiac disorders) | 3 (4)
Hypertension (Vascular disorders) | 2 (2)
Renal Complications (Renal and urinary disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Arteriovenous Fistula (Vascular disorders) | 1 (2)
Infection (non-sepsis) (Infections and infestations) | 2 (3)
Claudication (Non-target limb) (Vascular disorders) | 3 (4)
Claudication (Target Limb) (Vascular disorders) | 2 (2)
Dissection (Target Vessel) (Surgical and medical procedures) | 1 (1)
Critical Limb Ischemia (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Aneurysm (Site Other) (Vascular disorders) | 1 (1)
Cerebrovascular Disease (Nervous system disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Ischemic Colitis (Gastrointestinal disorders) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Myocardial Ischemia (Cardiac disorders) | 1 (1)
Prostatic Hypertrophy (Reproductive system and breast disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Valvular Heart Disease (Cardiac disorders) | 1 (1)
Cardiovascular Disease (Cardiac disorders) | 1 (1)
Squamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arterial Perforation/Rupture (Vascular disorders) | 1 (1)
Revascularization Target Limb (Surgical and medical procedures) | 1 (1)
Upper Extremity Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luminexx Iliac Stent and Delivery System (N=134)
Pain (General disorders) | 6 (8)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Angina/Coronary Ischemia (Cardiac disorders) | 2 (2)
Bleeding (Vascular disorders) | 2 (2)
Renal Complications (Renal and urinary disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less